CLINICAL TRIAL: NCT04929067
Title: Immunotherapy Combined With Neoadjuvant Chemotherapy in Patients With Locally Advanced HPV (-) Head and Neck Squamous Cell Carcinoma
Brief Title: Efficacy and Safety of Immunotherapy Combined With Neoadjuvant Chemotherapy in Patients With Locally Advanced HPV (-) Head and Neck Squamous Cell Carcinoma: a Phase II Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhejiang University
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Efficacy and Safety of Immunotherapy Combined With Neoadjuvant Chemotherapy in Patients With Locally Advanced HPV (-) HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy combined with neoadjuvant chemotherapy forlocally advanced HNSCC (Experimental)
  Interventions: Drug: immunotherapy combined with neoadjuvant chemotherapy in patients with locally advanced HPV (-) head and neck squamous cell carcinoma

INTERVENTIONS:
Drug: immunotherapy combined with neoadjuvant chemotherapy in patients with locally advanced HPV (-) head and neck squamous cell carcinoma — immunotherapy combined with neoadjuvant chemotherapy in patients with locally advanced HPV (-) head and neck squamous cell carcinoma

SUMMARY:
There are few clinical trials of chemotherapy combined with immunotherapy in the neoadjuvant stage of locally advanced head and neck squamous cell carcinoma. The "phase II clinical trial of efficacy and safety of immunotherapy combined with neoadjuvant chemotherapy in patients with locally advanced HPV (-) head and neck squamous cell carcinoma" carried out by our team will be an active exploration of the application of immunodrugs in the neoadjuvant stage of newly treated patients with locally advanced head and neck squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria: 1. The patients voluntarily participated in the clinical trial and signed the informed consent; 2. Histologically and pathologically confirmed locally advanced (stage Ⅲ - Ⅳ b) and HPV (-) head and neck squamous cell carcinoma. The primary tumor sites included oral cavity, oropharynx, larynx and hypopharynx; 3. The newly diagnosed patients did not receive any anti-tumor treatment ; 4. At least one measurable lesion (RECIST v1.1); 5. PS score was 0-1; 6. The main organ function met the following criteria within 7 days before treatment ① Blood routine examination standard (without blood transfusion within 14 days) Hemoglobin (HB) ≥ 90g / L; Absolute neutrophil count (ANC) ≥ 1.5 × 10*9/L；Platelet count (PLT) ≥ 80 × 10*9/L；② Biochemical test standard: Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN; Serum creatinine (CR) ≤ 1.5 ULN or creatinine clearance rate (CCR) ≥ 60 ml / min; ③ Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%); 7. Women of childbearing age should agree to use contraceptive measures (such as intrauterine device, contraceptive or condom) during the study period and within 6 months after the end of the study; Serum or urine pregnancy test was negative within 7 days before study enrollment. Male patients should agree to use contraception during the study period and within 6 months after the end of the study period.

-

Exclusion Criteria: 1) Patients with carcinoma of nasal cavity and paranasal sinuses, nasopharyngeal carcinoma and HPV (+) oropharyngeal carcinoma;

2) Patients who have used immune checkpoint inhibitors (including PD-1, PD-L1, PD-L2 and CTLA-4 inhibitors) in the past;

3) At the same time, there were other malignant tumors which were not controlled or under treatment;

4) Patients with any severe and / or uncontrolled medical disease include:

* The patients who used at least two kinds of antihypertensive drugs still had poor blood pressure control (systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg);

  * Grade 1 or above myocardial ischemia or myocardial infarction and grade 2 or above congestive heart failure (NYHA classification);

    * Sinus bradycardia; Or second degree or more atrioventricular block, or sinus arrest (except pacemaker installed); Arrhythmia (including QTc ≥ 480ms); It is necessary to use drugs known to prolong QTc interval, including antiarrhythmic therapy;

      * Active or uncontrolled severe infection (≥ CTC AE grade 2 infection);

        * Patients with liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need antiviral drugs;

          ⑥ Renal failure requiring hemodialysis or peritoneal dialysis;

          ⑦ History of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or organ transplantation;

          ⑧ The patients with diabetes had poor blood glucose control (FBG > 10mmol / L);
          * Urine routine examination showed that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0g;

            5) Patients who received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment;

            6) The imaging findings showed that the tumor formed deep ulcer, or had invaded important blood vessels, or the researchers judged that fatal massive hemorrhage might occur during the follow-up study;

            7) Regardless of the severity, there are any signs or history of bleeding constitution; In the first 4 weeks, there was any bleeding or bleeding event ≥ CTC AE 3; There are unhealed wounds, ulcers or fractures;

            8) In the first 6 months of the study, patients with arteriovenous thrombotic events such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism occurred;

            9) Patients with history of aneurysm / dissection;

            10) Patients with history of epilepsy or ataxia of nervous system need treatment;

            11) Those who have a history of psychotropic drug abuse and can't quit or have mental disorder;

            12) Patients with history of peripheral nervous system diseases and muscle strength below grade 3;

            13) Those who had participated in other anti-tumor drug clinical trials or were conducting other clinical trials within 4 weeks before enrollment;

            14) They can not tolerate the drugs used in this project, including treprizumab, albumin, paclitaxel and cisplatin, or have a history of severe hypersensitivity to any component;

            15) According to the judgment of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response rate for participants after receiving immunotherapy combined with neoadjuvant chemotherapy | 5 year

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 year
Major pathological response rate for the patients who received radical surgery | 5 year
Progression free survival | 5 year
Overall survival | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No